CLINICAL TRIAL: NCT04132375
Title: A Double-blind, Placebo-controlled, Adaptive, Phase 2/3 Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of INM004 in Pediatric Patients With Shiga Toxin-positive Bloody Diarrhea for Prevention of Hemolytic Uremic Syndrome
Brief Title: Phase 2/3 Study to Evaluate PK, Safety & Efficacy of INM004 in STEC Positive Pediatric Patients for Prevention of HUS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to COVID pandemia enrolment was stopped on 20March2020
Sponsor: Inmunova S.A. (Other)
Collaborators: Exeltis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-INM004-02
Record Dates: First submitted 2019-07-19; First posted 2019-10-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-03

CONDITIONS: Bloody Diarrhea; STEC, Unspecified; Hemolytic-Uremic Syndrome; Pediatric Kidney Disease
MeSH Terms: conditions — Hemolytic-Uremic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will be an adaptive seamless design (ASD) phase 2/3 investigation using an "inferentially seamless" platform.
  Stage 1 In Stage 1, subjects will be randomly assigned to receive 1 of the 3 treatment regimens (high treatment regimen, low treatment regimen, or placebo) in a 1:1:1 ratio.
  Review for Dose Selection The Data Monitoring Committee will conduct a blinded safety review at the end of Stage 1 to determine the best active dose based on safety.
  Stage 2 Stage 2 is considered the efficacy portion of the study. The randomization ratio for subjects in Stage 2 will be 1:1 (active treatment regimen of INM004: placebo).
  Interim Analysis The intent of the unblinded interim analysis is to demonstrate superiority of INM004 versus the placebo, based on 80% reduction in the incidence of HUS in the treated cohort to stop study due to overwhelming efficacy, or declare futility, or re-estimate sample.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Double-blind, Placebo-controlled, IWRS based. access to unblinded interim results will be limited to the DMC and unblinded statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stage 1 - high treatment arm (Active Comparator): Subjects will receive a 1st intravenous dose of 4 mg/kg INM004 (Anti-Stx hyperimmune equine immunoglobulin F[ab']2 fragments) and a 2nd intravenous dose of 4 mg/kg of INM004. Each dose will be separated by 24 h (± 2 h).
  Interventions: Drug: INM004
- Stage 1 - Low treatment arm (Active Comparator): Subjects will receive a 1st intravenous dose of 4 mg/kg INM004 (Anti-Stx hyperimmune equine immunoglobulin F[ab']2 fragments) and a 2nd intravenous dose of Placebo. Each dose will be separated by 24 h (± 2 h).
  Interventions: Drug: INM004
- Stage 1 - Placebo arm (Placebo Comparator): Subjects will receive a 1st intravenous dose of Placebo and a 2nd intravenous dose of Placebo. Each dose will be separated by 24 h (± 2 h).
  Interventions: Drug: Placebo
- Stage 2 - Selected active treatment arm (Active Comparator): In the case, the high treatment regime is selected, subjects will receive a 1st intravenous dose of 4 mg/kg INM004 and a 2nd intravenous dose of 4 mg/kg of INM004. Each dose will be separated by 24 h (± 2 h).
  In the case, the low treatment regime is selected subjects will receive an intravenous dose of 4 mg/kg INM004
  Interventions: Drug: INM004
- Stage 2 - Placebo arm (Active Comparator): In the case, the high treatment regime is selected, subjects will receive a 1st intravenous dose of Placebo and a 2nd intravenous dose of Placebo, each dose separated by 24 h (± 2 h)
  In the case, low treatment regime is selected subjects will receive a single intravenous dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INM004 — The IMP dose to be studied will be 4 mg of protein/kg of subject's weight. Each vial contains 25 mg protein/mL. Therefore, each subject must receive 0.16 mL/kg.
  The IMP will be added to the 100 mL infusion bag of saline solution. Doses will be administered as an infusion at 2.0 mL/min over 50 min with an interval of 24 h between doses.
  Other Names: active
  Arms: Stage 1 - Low treatment arm; Stage 1 - high treatment arm; Stage 2 - Selected active treatment arm
Drug: Placebo — The IMP dose to be studied will be 4 mg of protein/kg of subject's weight. Each vial contains 25 mg protein/mL. Therefore, each subject must receive 0.16 mL/kg.
  The IMP will be added to the 100 mL infusion bag of saline solution. Doses will be administered as an infusion at 2.0 mL/min over 50 min with an interval of 24 h between doses.
  Arms: Stage 1 - Placebo arm; Stage 2 - Placebo arm

SUMMARY:
The investigational medicinal product (IMP), INM004, proposes to neutralize the toxin in the bloodstream to prevent the interaction of the Stx with the specific receptor, by means of a polyclonal antibody to be administered upon the appearance of symptoms (bloody diarrhea) and diagnosis of infection by STEC, thereby preventing the action of the toxin in the body. Thus, the initial hypothesis for examination is for the prevention of the full expression of HUS, based upon presumptive clinical, biochemical, and other biological evidence suggesting a risk of HUS at the time of treatment application. The polyclonal antibody (F(ab')2 fragment) is obtained by processing the serum of equine animals previously immunized against engineered Stx1B and Stx2B immunogens.

INM004 could be administered at the earlier stages of STEC disease since subjects with STEC diarrhea are more likely to benefit from Stx neutralizing antibodies before the development of extra-intestinal manifestations and HUS. Neutralizing equine anti-Stx F(ab')2 antibodies (INM004) have the objective of preventing the development of HUS by blocking the circulating toxins in patients infected with STEC. Therefore, INM004 may be used in patients with a clinical manifestation of bloody diarrhea and a positive Stx result in feces. Early interruption of the Stx mediated cascade is expected to prevent the development of HUS, alleviate the severity of the illness, the rate of complications and the incidence/duration of hospitalizations. Therefore, patients in the early phases of the disease will be targeted in this study, ie, children who seek medical care due to diarrhea associated with STEC infection before HUS development.

DETAILED DESCRIPTION:
Hemolytic uremic syndrome (HUS) is a form of thrombotic microangiopathy, characterized by microangiopathic hemolytic anemia, thrombocytopenia, and acute renal impairment of varying severity, which may be preceded by an episode of diarrhea with or without blood. Karmali et al. showed the relationship between this syndrome and diarrhea caused by Shiga toxin-producing bacteria such as Escherichia coli. These cytotoxins, called Shiga-like toxins or Shiga toxins (Stx), are also called verotoxins, due to the characteristic cytopathic effect they cause on Vero cell cultures.

HUS is often classified into 3 primary types: 1) HUS due to infections associated with Shiga-toxin producing E. coli (STEC) or Shigella dysenteriae Type 1, often associated with diarrhea, with the rare exception of HUS due to a severe disseminated infection caused by Streptococcus pneumoniae, 2) HUS related to complement abnormalities or related to factor ADAMTS13 deficit, such HUS is also known as "atypical HUS" and is not associated with diarrhea, and 3) HUS of unknown etiology that usually occurs in the course of systemic diseases or physio-pathologic conditions such as pregnancy, after transplantation or after drug use.

E. coli bacteria normally live in the intestines of people and animals. Cattle and sheep are the main reservoirs of STEC, and the major transmission route is believed to be food contaminated with animal feces. Contaminated water has also been recognized as a source, and direct human-to-human and animal-to-human transmission have been reported.

E. coli consists of a diverse group of bacteria. Most of them are harmless and an important part of a healthy human intestinal tract. However, some E. coli are pathogenic, that can cause either diarrhea or illness outside of the intestinal tract. Diarrheagenic E. coli strains are categorized into 6 pathotypes: 1) Enterotoxigenic E. coli, 2) Enteropathogenic E. coli, 3) Enteroaggregative E. coli, 4) Enteroinvasive E. coli, 5) diffusely adherent E. coli, and 6) STEC. STEC may also be referred to as verocytotoxin-producing E. coli (VTEC). This last pathotype is the one most commonly associated with foodborne outbreaks.

Treatment of STEC HUS renal damage caused by Stx is available. The investigational medicinal product (IMP), INM004, proposes to neutralize the toxin in the bloodstream to prevent the interaction of the Stx with the specific receptor, by means of a polyclonal antibody to be administered upon the appearance of symptoms (bloody diarrhea) and diagnosis of infection by STEC, thereby preventing the action of the toxin in the body. Thus, the initial hypothesis for examination is for the prevention of the full expression of HUS, based upon presumptive clinical, biochemical, and other biological evidence suggesting a risk of HUS at the time of treatment application. The polyclonal antibody (F(ab')2 fragment) is obtained by processing the serum of equine animals previously immunized against engineered Stx1B and Stx2B immunogens.

INM004 could be administered at the earlier stages of STEC disease since subjects with STEC diarrhea are more likely to benefit from Stx neutralizing antibodies before the development of extra-intestinal manifestations and HUS. Neutralizing equine anti-Stx F(ab')2 antibodies (INM004) have the objective of preventing the development of HUS by blocking the circulating toxins in patients infected with STEC. Therefore, INM004 may be used in patients with a clinical manifestation of bloody diarrhea and a positive Stx result in feces. Early interruption of the Stx mediated cascade is expected to prevent the development of HUS, alleviate the severity of the illness, the rate of complications and the incidence/duration of hospitalizations. Therefore, patients in the early phases of the disease will be targeted in this study, ie, children who seek medical care due to diarrhea associated with STEC infection before HUS development.

Pediatric subjects between 1 and 10 years (y) of age at the time of screening with an increased risk for development of HUS defined by the presence of bloody diarrhea based upon history or presentation and positive screen for Stx2 in the stool will be enrolled.

Bloody diarrhea and positive screen for Stx2 have been included as inclusion criteria as these factors have been identified as risk factor for HUS development and will serve to enrich the patient population within the study to those most likely to benefit from this therapy.

Case of Bloody Diarrhea Any person with an increase in the number of daily stools and alteration in the stool consistency, with presence of visible blood, which may include episodes of stool formed with blood in the form of streaks on its surface or blood visible only under a microscope, which may be accompanied by other symptoms such as vomiting, nausea, abdominal pain, or fever.

Case of Shiga Toxin producing Escherichia coli Infection

Identification of the etiological agent by at least 1 of the following laboratory criteria:

* Isolation of an E. coli strain that produces Stx or harbors stx1 or stx2 gene(s);
* Direct detection of stx1 or stx2 gene(s) nucleic acid (without strain isolation);
* Direct detection of free Stx in feces (without strain isolation). The surveillance of the STEC strains is performed using subtyping techniques: 1) genotyping of stx and eae by polymerase chain reaction (PCR)-restriction fragment length polymorphism and 2) pulsed-field gel electrophoresis. STEC O157 and non O157 strains are recovered from the clinic, animal, food and environmental samples, and E. coli O157:H7, a Stx2a/Stx2c producer, harboring eae and ehxA genes, is the most common serotype.

Case of Hemolytic Uremic Syndrome Patient of any age who presents in an acute form with microangiopathic hemolytic anemia, thrombocytopenia, and renal compromise.

Case of Hemolytic Uremic Syndrome with Confirmed Diagnosis of Shiga Toxin producing Escherichia coli

Case of HUS with identification of the etiological agent by at least 1 of the laboratory criteria:

* Screening of stx1 and/or stx2 by PCR/isolation of STEC
* Detection of free Stx in stool
* Detection of serogroup-specific O antigen antibodies O157, O145, O121

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 1 to < 10 y.
2. Signed informed consent from the parent(s)/legal guardian with assent from the subject as appropriate by age and regulatory guidance.
3. Bloody diarrhea based upon history or presentation (by visual inspection).
4. Detection of Stx2 in stool based on enzyme immunoassay (EIA) and/or stx2 based on PCR before randomization.

   NOTE: The basis for accepting a positive test for stx2 by EIA is based on taking as valid the results yielded from an EIA whose sensitivity and specificity are greater than 98.7% and 100%, respectively (according to the description in the insert) as per recommendation given by the NRL. The Sponsor will select the investigational sites that have in their laboratory such EIA test used in the STEC diagnostic routine algorithm. (Appendix 6).
5. For children between 1 to 5 years old: weight for length/height between percentiles 3 (< 2 z score) and 97 (> 2 z score) corresponding to age (according to the reference tables "WHO Child Growth Standards".
6. For children ≥ 5 years: Body mass index (BMI) between percentiles 3 (<2 z score) and 97 (> 2 z score) corresponding to age (according to the reference tables "WHO Child Standards, Appendix 4)

Exclusion Criteria:

1. Any laboratory findings compatible with the development of HUS:

   * Microangiopathic hemolytic anemia defined as LDH above the ULN for age with the finding of schistocytes on peripheral smear and a negative Coomb's test, and/or
   * Thrombocytopenia: platelet count < 150 × 103/μL, and/or
   * Renal failure: serum creatinine > ULN adjusted for age and gender criteria despite correction of hypovolemia, and/or hematuria, and/or proteinuria (Table 7.1)11 NOTE: Laboratory results must be obtained within 24 h before the 1st study drug administration; there must be no clinical signs and symptoms of HUS at the time laboratory assessments are obtained. If there is any change in clinical presentation in the 24 h before the 1st study drug administration, laboratory assessments are to be repeated and results reviewed before study drug administration.

   NOTE: Laboratory and physical examination results must indicate normal hydration before the 1st study drug administration.
2. A history of chronic/recurrent hemolytic anemia, thrombocytopenia, or chronic renal failure.
3. A family history of aHUS.
4. Anuria or oliguria after hypovolemia is corrected.
5. Evidence of clinically significant chronic active disease not medically controlled.
6. History of anaphylaxis, prior administration of equine serum (eg, antitetanus serum or anti-ophidic serum, or anti-arachnid toxin serum), or allergic reaction to contact with, or exposure to, horses.
7. Family relation or work relation with a member of the personnel of the research group.

   -

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Incidence of HUS development | 4 weeks
  The primary endpoint is a binary (Y/N) endpoint defined as having confirmed HUS by week 4. This endpoint will be centrally adjudicated by a Clinical Endpoint Committee. This committee will classify all potential events into one of the following categories:
  * Confirmed HUS
  * Probable HUS
  * No HUS
  The proportion of children with HUS by week 4 confirmed by central adjudication will be reported for each treatment arm (optimal dose of INM004 vs placebo).

SECONDARY OUTCOMES:
Frequency of subjects with treatment-emergent adverse event (TEAEs) to assess the safety of 2 doses of INM004 in children through evaluation of safety data in Stage 1 | 12 weeks
  Frequency of subjects with TEAEs will be summarized by treatment group providing the number of subjects with event, the proportion subjects with event and the number of events
  The statistics above will also be provided for the following events:
  * Serious TEAEs
  * TEAEs leading to study withdrawal
  * Treatment related TEAEs
  * Serious and treatment related TEAEs
  * Severe TEAEs
  * TEAEs leading to death
  * treatment emergent adverse events of special interest (TEAESI)
  * treatment-emergent adverse events related to background disease (TEAEBD) The frequency of TEAEs will also be reported by System Organ Class (SOC), and will also be reported by severity and relationship to study drug.
  AEs will be coded by Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) classification
Frequency of subjects with treatment-emergent adverse event (TEAEs) to assess the safety of the administration on INM004 in all treated patients | 12 weeks
  Frequency of subjects with TEAEs will be summarized by treatment group providing the number of subjects with event, the proportion subjects with event and the number of events
  The statistics above will also be provided for the following events:
  * Serious TEAEs
  * TEAEs leading to study withdrawal
  * Treatment related TEAEs
  * Serious and treatment related TEAEs
  * Severe TEAEs
  * TEAEs leading to death
  * treatment emergent adverse events of special interest (TEAESI)
  * treatment-emergent adverse events related to background disease (TEAEBD) The frequency of TEAEs will also be reported by System Organ Class (SOC), and will also be reported by severity and relationship to study drug.
  AEs will be coded by Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) classification
Incidence of secondary endpoints through Week 4 and Week 12 (short term complications). | by Week 4; by Week 12
  * the time to death will be calculated in order to assess overall survival,
  * The time to the first serious extrarenal events will be calculated (in days) for the following events:
    * Major neurological involvement
    * Cardiovascular involvement
    * Gastrointestinal involvement
    * Pancreatic involvement
    * Hepatic involvement
Incidence in long-term sequelae from Week 12 through Week 48 in those who develop HUS (long-term complications). | From Week 12 through Week 48
  The time to long-term sequelae will be calculated for the following events:
  * Long-term renal sequelae
  * Neurological sequelae
  * Cardiovascular sequelae
  * Pancreatic sequelae
  * Gastrointestinal sequelae
  * Overall survival
Time after the administration of INM004 in which peak plasma concentration is reached (Tmax) | 5 days
  Pharmacokinetic profile will be assessed by measuring serum INM004 concentration at different timepoints. Serum INM004 concentration will be followed by a specific ELISA. Concentration of INM004 will be plotted as a function of time and pharmacokinetic profile will be defined.
Peak Plasma Concentration (Cmax) of INM004 | 5 days
  Pharmacokinetic profile will be assessed by measuring serum INM004 concentration at different timepoints. Serum INM004 concentration will be followed by a specific ELISA. Concentration of INM004 will be plotted as a function of time and pharmacokinetic profile will be defined.
Area under the plasma concentration of INM004 versus time curve (AUC) | 5 days
  Pharmacokinetic profile will be assessed by measuring serum INM004 concentration at different timepoints. Serum INM004 concentration will be followed by a specific ELISA. Concentration of INM004 will be plotted as a function of time and pharmacokinetic profile will be defined.

OTHER OUTCOMES:
Length of the hospital stay in subjects who developed HUS | 4 weeks
  Length of the hospital stay will be calculated as the discharge date minus the admission date + 1 as collected in the HUS admission/ discharge forms .
Other observed or derived estimates of staff and resource utilization in subjects who developed HUS | 4 weeks
  The following resources, measured in duration of days, utilized during the entire hospitalization for HUS will be collected: peritoneal dialysis, hemodialysis, transfusions, antibiotics, erythropoietin, plasmapheresis, diuretics, frozen plasma, hypotensors, mechanical ventilation, insulin duration in the intensive care unit, duration in the general ward and abdominal surgery
Incidence of predictors of mortality in subjects who developed HUS. | 4 weeks
  For each subject hospitalized for HUS, the following binary (Y/N) variables will be created:
  * White blood cell (WBC) value > 20,000/mL
  * Hemoglobin (Hb) value > 10.8 g/dL
  * Sodium (Na) < 128 mEq/L
  * Neurological involvement
Serotype and genotype of E. coli strains isolated from all subjects | 4 weeks
  All E. coli strains isolated from patients will be Serotyped and genotyped. A correlation between a certain type of strain and the development of HUS will be investigated. Strains will be aggregated by serotype and/or genotype and a correlation between a specific combination and development of HUS will be explored.
Changes from baseline in laboratory parameters following study drug administration in all subjects. | 4 weeks
  Descriptive statistics will be produced for the values and the changes from baseline at each assessment time point by treatment arm.
  The absolute frequency (n) and percentage (%) of subjects with clinically significant abnormalities by visit and at any post-baseline moment during the study will be reported by treatment arm.
immunogenicity of INM004 by measuring anti-INM004 antibodies at day 30 post drug administration. | 4 weeks
  Assessment of the immunogenicity of INM004 determined by the presence of anti-drug antibodies (ADA) in serum samples by a specific ELISA test. This will be evaluated at baseline and at day 30 post drug administration
Investigator submitted events (ie, confirmed HUS, incomplete HUS, or signs and symptoms which may represent neither) for hypothesis generation. | 4 weeks
  * A secondary binary endpoint defined as having either probable or confirmed HUS by week 4 will be defined using the CEC assessment.
  * A secondary qualitative endpoint defined as having either mild, moderate or severe HUS (probable or confirmed) by week 4 will be defined using the CEC assessment.

CONTACTS AND LOCATIONS:
Overall Officials: SANTIAGO SANGUINETI, PhD, Study Director — Inmunova S.A.
Locations (7):
- Argentina (7):
  - Hospital Penna, Bahía Blanca, Buenos Aires
  - Hospital Sor Maria Ludovica, La Plata, Buenos Aires
  - Hospital Lucio Molas, Santa Rosa, La Pampa Province
  - Hospital Castro Rendon, Neuquén, Neuquén Province
  - Hospital Elizalde, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Hospital Orlando Alassia, Santa Fe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Imdad A, Mackoff SP, Urciuoli DM, Syed T, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD012997. doi: 10.1002/14651858.CD012997.pub2. PMID 34219224